CLINICAL TRIAL: NCT02703402
Title: Effects of an Exercise Program Under Supervision and Unsupervised in the Treatment of Low Back Pain: a Randomized Clinical Trial
Brief Title: Effects of an Exercise Program Under Supervision and Unsupervised in the Treatment of Low Back
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0526
Record Dates: First submitted 2016-02-17; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Low Back Pain
Keywords: low back pain; physical exercise and quality of life
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise protocol (Experimental): Will complete all the protocol of exercises with orientation and attendance directly from a professional of physical education, in the Service of Physiatry and Rehabilitation in HCPA
  Interventions: Other: Exercise protocol
- Manual of exercises (Experimental): Treatment Group: will complete one session of the protocol of exercises with orientation and attendance directly from a professional of Physical Education, in the service of Physiatry and Rehabilitation of HCPA, to clarify any doubts about the protocol. The further sessions will be completed at home, along weekly monitoring of the researchers through phone calls, the patients of this group will receive a manual with the sequence of the exercises.
  Interventions: Other: Manual of exercises

INTERVENTIONS:
Other: Exercise protocol — Control group will complete all the protocol of exercises with orientation and attendance directly from a professional of physical education, in the Service of Physiatry and Rehabilitation in HCPA.
  Arms: Exercise protocol
Other: Manual of exercises — Treatment group will complete one session of the protocol of exercises with orientation and attendance directly from a professional of Physical Education, in the service of Physiatry and Rehabilitation of HCPA, to clarify any doubts about the protocol. The further sessions will be completed at home, along weekly monitoring of the researchers through phone calls, the patients of this group will receive a manual with the sequence of the exercises
  Arms: Manual of exercises

SUMMARY:
ABSTRACT: Low back pain is one of the most frequent causes of incapacity. The prevalence of this syndrome is 60-85% for the survival of the individuals. Among the most promising strategies of low back pain intervention, is the physical activity that is usually associated with a long list of health benefits.

DETAILED DESCRIPTION:
Purpose: evaluate the efficacy of a protocol of exercises to low back pain rehabilitation under supervision of physiatry service and rehabilitation in the Hospital de Clínicas de Porto Alegre compared with same protocol performed at home in regards to pain.

Methods: Randomized clinical trial with a sample of 122 subjects of the community of both sex, with ages between 30 to 55, with low back pain complain. These subjects will accomplish during 12 weeks protocol of exercises from "Exercises to low back pain" Physiatry and Rehabilitation service from HCPA, randomized in two groups: group 1 will complete all the protocol of exercises with orientation and attendance directly from a professional of physical education, in the Service of Physiatry and Rehabilitation in HCPA. Group 2 will complete one session of the protocol of exercises with orientation and attendance directly from a professional of Physical Education, in the service of Physiatry and Rehabilitation of HCPA, to clarify any doubts about the protocol. The further sessions will be completed at home, along weekly monitoring of the researchers through phone calls, the patients of this group will receive a manual with the sequence of the exercises.

ELIGIBILITY:
Inclusion Criteria:

* ages between 30 and 55
* Pain should be without radiation to lower body
* Pain with more than 12 weeks of evolution.
* Visual Analog Scale of Pain (VAS) should present a pattern above 3 (moderate).

Exclusion Criteria:

* Patients with Exclusion Criteria: will be excluded those patients that present musculoskeletal impairment in lower body,
* After surgery and anesthetic block.
* individuals affected with comorbidities
* Patients with rheumatic diseases, recent fractures, tumors, pregnant women, smokers and general practitioners of physical activity.
* Subjects who are unable to attend the hospital twice a week.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Pain Scale to asses Low Back Pain | 24 months
  Visual Analogue Pain Scale (EVA) - change from baseline pain after the intervention - evaluates the intensity of pain using a ruler divided into eleven equal parts, with a classification from 0 (painless) and 10 (maximum pain).

SECONDARY OUTCOMES:
Short-Form Survey (SF-36) to evaluate life quality | 24 months
  change from baseline in life quality after intervention -Survey with 36 items that measure 8 variable.
Six minutes walk-test - Functional capacity | 24 months
  Change from baseline in functional capacity ater intervention - measure the distance walked during 6 minutes. Performed in a corridor with a 30 meter distance with two cones in the extremities.
sit and reach test - flexibility | 24 months
  change from baseline in flexibility after intervention - individual in the sitting position with legs extended oriented move the marker on millimeter surface, held 3 times and considered the greatest value

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C. dos Santos, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ben Salah Frih Z, Fendri Y, Jellad A, Boudoukhane S, Rejeb N. Efficacy and treatment compliance of a home-based rehabilitation programme for chronic low back pain: a randomized, controlled study. Ann Phys Rehabil Med. 2009 Jul;52(6):485-96. doi: 10.1016/j.rehab.2009.04.002. Epub 2009 May 15. English, French. PMID 19473905
- [Background] Descarreaux M, Normand MC, Laurencelle L, Dugas C. Evaluation of a specific home exercise program for low back pain. J Manipulative Physiol Ther. 2002 Oct;25(8):497-503. doi: 10.1067/mmt.2002.127078. PMID 12381971
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Hartvigsen J, Morso L, Bendix T, Manniche C. Supervised and non-supervised Nordic walking in the treatment of chronic low back pain: a single blind randomized clinical trial. BMC Musculoskelet Disord. 2010 Feb 10;11:30. doi: 10.1186/1471-2474-11-30. PMID 20146793
- [Background] Brown CA. The beliefs of people with chronic pain in relation to 'important' treatment components. Eur J Pain. 2004 Aug;8(4):325-33. doi: 10.1016/j.ejpain.2003.10.005. PMID 15207513
- [Background] Shirado O, Doi T, Akai M, Hoshino Y, Fujino K, Hayashi K, Marui E, Iwaya T; Japan Low back-pain Exercise Therapy Study; Investigators Japanese Orthopaedic Association; Japanese Society for Musculoskeletal Rehabilitation; Japanese Clinical Orthopaedic Association. Multicenter randomized controlled trial to evaluate the effect of home-based exercise on patients with chronic low back pain: the Japan low back pain exercise therapy study. Spine (Phila Pa 1976). 2010 Aug 1;35(17):E811-9. doi: 10.1097/BRS.0b013e3181d7a4d2. PMID 20628332
- [Background] Kuukkanen T, Malkia E, Kautiainen H, Pohjolainen T. Effectiveness of a home exercise programme in low back pain: a randomized five-year follow-up study. Physiother Res Int. 2007 Dec;12(4):213-24. doi: 10.1002/pri.378. PMID 17849435
- [Background] Vuori IM. Dose-response of physical activity and low back pain, osteoarthritis, and osteoporosis. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S551-86; discussion 609-10. doi: 10.1097/00005768-200106001-00026. PMID 11427782
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180